CLINICAL TRIAL: NCT05973396
Title: The Effects of Mental and Physical Fatigue to Force Production in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PUIRB-2022-11
Record Dates: First submitted 2022-11-08; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Mental Fatigue; Muscle Weakness
Keywords: Force Production; Muscular Fatigue; Mental Cognition
MeSH Terms: conditions — Mental Fatigue; Muscle Weakness | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Physical Fatigue only (Active Comparator): Rogue Echo Bike 20 intervals of 10 second of maximal-submaximal effort to 50 seconds of recovery low intensity effort
  Interventions: Other: Physical Fatiguing Task only
- Experiment: Mental and Physical Fatigue (Experimental): Rogue Echo Bike 20 intervals of 10 second of maximal-submaximal effort to 50 seconds of recovery low intensity effort with mentally fatiguing task during low intensity effort pace with stroop testing during 50 seconds
  Interventions: Other: Physical and Mental Fatiguing Task

INTERVENTIONS:
Other: Physical Fatiguing Task only — Control group: 20-25 minutes [Rogue Echo Bike 20 intervals of 10 second of maximal-submaximal effort to 50 seconds of recovery low intensity effort] without mentally fatiguing task during low intensity effort pace
  Other Names: Physical and Mental Fatiguing Task
  Arms: Control: Physical Fatigue only
Other: Physical and Mental Fatiguing Task — Experimental group: 20-25 minutes [Rogue Echo Bike 20 intervals of 10 second of maximal-submaximal effort to 50 seconds of recovery low intensity effort] with mentally fatiguing task during low intensity effort pace (which includes: stroop test)
  Arms: Experiment: Mental and Physical Fatigue

SUMMARY:
The primary objective is to investigate the correlation between physical and mental fatigue to lower extremity force production in adults to determine if there is an association of performance output that is inhibited by mental and physical stressors that mimic sport environments that can be further investigated to determine the importance of not only physical training and exercise for athletes, but also mental and cognitive exercises with physical task to enhance performance training and rehabilitation of individuals.

In adults, how does physical and mental fatigue in combination compared to those who are just physically fatigued affect average peak height in performance of five CMJ with hands on hips.

DETAILED DESCRIPTION:
In terms of injury prevention mental or cognitive fatigue and altered biomechanics play a large role in risk of injury or reinjury. This can lead to disturbances in gait, balance or even It is known that there are decreases in rate of force production in a physically fatigued state.

However, this does not show if a mentally fatigued and physically fatigued individual have any negative implications towards a more dynamic and reactive test and conditions that mimic sport more than static balancing or linear walking. It is even noted in reactive times of post ACLr (one of the most common sports related injuries) have lower reactive times in agility test With ACLr having a high level or rate or reinjury on surgical side and nonsurgical side as well as known alterations of the cerebellum and specifically the primary sensory cortex.Understanding how much a mental and physical fatigue can impact reactive cognition and force production can be vital key in not only sports performance and management, but also risk or injury and be associated in the plan of returning an athlete to sport as power and force production is a key determinant of performance in many individual and team sports. It is noted that physical activities directly enhance mental fatigue significantly, but it is widely unresearched objectively how much or when physical fatigue directly impacts mental cognition and decision making properties to an individual. In sport it is crucial to act and react to be able to be successful. Multidirectional and team sports involve constant mental cognition in terms of visual, auditory interpretation and cognition, ability to recognize patterns and to finally physically perform tasks in a highly efficient manner.

The goal of an athlete is to be conditioned to play their best whether that is the first minute of the game or its last. That means making the correct decision and physically performing it. However, in a fatigued state can the athlete properly perform what is needed to be done in a safe and effective manner that is comparable to a not fatigued state.

ELIGIBILITY:
Inclusion Criteria:

Current students at Parker University from the ages of 21 to 65 years for safety concerns Children were not considered for this study Elderly were not considered for this study Current students who are currently physically active at least once a week

Exclusion Criteria:

1. Anyone with who self reports previous history of cardiovascular issues or hospitalizations Rationale: Participants will be doing aerobic/ anaerobic efforts that will increase their heart rate Source: Redcap Questionnaire, Baseline visit
2. Lower extremity surgery within the last two years Rationale: Puts participant more at risk of injury since inducing fatigue and a maximal power effort Source: Redcap Questionnaire, Baseline visit
3. Medical restrictions for full activity Rationale: Puts participant more at risk of injury since inducing fatigue and a maximal power effort Source: Redcap Questionnaire, Baseline visit

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Average total height and force production of 5 Arms Fixed Countermovement jumps | 60 minutes
  Average total height and force production of 5 Arms Fixed Countermovement jumps

SECONDARY OUTCOMES:
Difference in mental math pre and post experiment scores | 60 minutes
  Difference in mental math pre and post experiment scores

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Pohlman, PhD, Study Director — Director of Research
Locations (2):
- United States (2):
  - ParkerFit, Dallas, Texas
  - Parker University, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.4085/1062-6050-266-18
- See also: Related Info — https://doi.org/10.1016/j.jsams.2018.07.004
- See also: Related Info — https://doi.org/10.3389/fneur.2018.00915
- See also: Related Info — https://doi.org/10.1007/s40279-013-0090-5